CLINICAL TRIAL: NCT00151177
Title: Feasibility and Efficacy Study of Early Continuous Positive Airway Pressure Ventilation in Patients With Acute Ischemic Stroke
Brief Title: Continuous Positive Airway Pressure Ventilation After Acute Ischemic Stroke
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Collaborators: New Health Sciences, Inc. (Industry); Rubel GmbH, Heiligenhaus, Germany (Unknown)
Responsible Party: Dr. M. Ritter, University_Hospital_Muenster
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMF-DZ-110413; NHSi2005-iCPAPAPNEASTROKE-001; UKM-SL-70234
Record Dates: First submitted 2005-09-07; First posted 2005-09-08 (Estimated); Last update posted 2010-11-24 (Estimated); Status verified 2008-04

CONDITIONS: Brain Infarction
Keywords: ischemic stroke; CPAP ventilation
MeSH Terms: conditions — Brain Infarction; Ischemic Stroke | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): treatment with three nights of CPAP ventilation starting the first night of admission
  Interventions: Device: non-invasive continuous positive airway pressure ventilation; Device: CPAP-treatment
- B (No Intervention): usual Stroke Unit care
  Interventions: Device: CPAP-treatment

INTERVENTIONS:
Device: non-invasive continuous positive airway pressure ventilation
  Arms: A
Device: CPAP-treatment — night time CPAP-mask ventilation

SUMMARY:
More than half of all stroke patients have sleep apneas in the acute phase after stroke. Sleep apneas may be associated with higher degrees of disability three months after stroke due to numerous factors associated with sleep apneas such as persistent hypertension, cardiac arrhythmias, and clotting disorders.

Non-invasive CPAP (continuous positive airway pressure)-therapy may reverse a number of these effects very shortly after initiation. The aim of the study is to test the feasibility of early non-invasive CPAP treatment starting in the first night after stroke onset, and to test its efficacy in a randomized clinical trial.

50 patients with acute ischemic stroke will be enrolled and randomly assigned to standard care PLUS CPAP treatment or standard care only. All patients randomized to the intervention group will receive CPAP therapy for the first three nights after stroke. In the fourth night, a cardiorespiratory polygraphy will be performed in patients and controls. Patients assigned to the intervention group with a respiratory distress index > 10/h will be treated further on. On admission, day 4, and day 10 after stroke, diffusion weighted MRI imaging will be performed to determine the size of the infarction. The NIHSS score will be used to assess clinical short-term outcome on day 4 and day 10. After three months, the outcome will be determined using the modified Rankin scale.

As CPAP therapy may be more laborious for the provider, the additional work-load will be documented using pre-specified scales.

Primary hypothesis of the study is, that CPAP therapy is feasible in acute stroke patients and that the additional work load will not outweigh the benefits.

Secondary hypothesis is that patients assigned to the treatment group have smaller infarctions on MRI and less neurological deficits at 3 months after stroke.

Patients entering the study will be investigated by transcranial Doppler ultrasound in case they have sufficient temporal bone windows for insonation and no stenosis or occlusions of major brain supplying arteries by the time of investigation that disturb the intracerebral blood flow.

All intracranial arteries will be assessed before treatment, after treatment and on day 8 after the insult.

Screen shots will be taken and will be analysed by dynamic vascular ultrasound (DVA), a new software algorithm developed by NHSi, to investigate microcirculatory information from the flow spectra of the major intracranial arteries.

The data from this post-hoc analysis are compared with the data of the polysomnography and with treatment.

Primary hypothesis in this substudy is that DVA reliably identifies patients with sleep apnea on days one and four after stroke. Secondary hypothesis is that DVA can distinguish between treated patients and controls.

ELIGIBILITY:
Inclusion criteria:

* AGE 18-85 years,
* NIH-SS 2-20 points,
* NIH-SS subitem 1a <=1.

Exclusion criteria:

* Modified Rankin Scale Score >=2 on admission
* primary intubation,
* Congestive heart failure (NYHA >=3),
* respiratory insufficiency
* recurrent vomiting
* absence of gag reflex,
* participation in another RCT

for the ultrasound sub-study

* absence of temporal bone window for insonation
* stenosis or occlusion of major brain supplying arteries interfering with normal blood flow

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2005-04; Primary Completion 2008-01 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Primary endpoint is to test the feasibility of early non-invasive CPAP ventilation in acute stroke patients

SECONDARY OUTCOMES:
Size of brain infarction on diffusion weighted MRI imaging at day 10 after symptom onset
Disability measured by the modified Rankin scale after three months

CONTACTS AND LOCATIONS:
Overall Officials: Darius G Nabavi, MD, Principal Investigator — University Hospital Muenster
Locations (1):
- University_Hospital_Muenster, Münster, Germany

REFERENCES:
- [Background] Turkington PM, Bamford J, Wanklyn P, Elliott MW. Prevalence and predictors of upper airway obstruction in the first 24 hours after acute stroke. Stroke. 2002 Aug;33(8):2037-42. doi: 10.1161/01.str.0000023576.94311.27. PMID 12154259
- [Background] Bassetti C, Aldrich MS, Quint D. Sleep-disordered breathing in patients with acute supra- and infratentorial strokes. A prospective study of 39 patients. Stroke. 1997 Sep;28(9):1765-72. doi: 10.1161/01.str.28.9.1765. PMID 9303023
- [Background] Iranzo A, Santamaria J, Berenguer J, Sanchez M, Chamorro A. Prevalence and clinical importance of sleep apnea in the first night after cerebral infarction. Neurology. 2002 Mar 26;58(6):911-6. doi: 10.1212/wnl.58.6.911. PMID 11914407
- [Derived] Minnerup J, Ritter MA, Wersching H, Kemmling A, Okegwo A, Schmidt A, Schilling M, Ringelstein EB, Schabitz WR, Young P, Dziewas R. Continuous positive airway pressure ventilation for acute ischemic stroke: a randomized feasibility study. Stroke. 2012 Apr;43(4):1137-9. doi: 10.1161/STROKEAHA.111.637611. Epub 2011 Dec 22. PMID 22198979